CLINICAL TRIAL: NCT02144714
Title: A Randomised, Single-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability and Immunogenicity of Three Formulations of Adalimumab (SB5, EU Sourced Humira® and US Sourced Humira®) in Healthy Subjects
Brief Title: Pharmacokinetic, Safety, Tolerability and Immunogenicity Study of SB5 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SB5-G11-NHV; 2013-005332-15 (EudraCT Number)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2018-09-21 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- SB5 (Experimental): SB5, single dose of 40 mg via subcutaneous injection (study drug)
  Interventions: Biological: SB5; Biological: EU sourced Humira®
- EU sourced Humira® (Active Comparator): EU sourced Humira®, single dose of 40 mg via subcutaneous injection (reference drug)
  Interventions: Biological: SB5; Biological: US sourced Humira®
- US sourced Humira® (Active Comparator): US sourced Humira®, single dose of 40 mg via subcutaneous injection (reference drug)
  Interventions: Biological: EU sourced Humira®; Biological: US sourced Humira®

INTERVENTIONS:
Biological: SB5
  Arms: EU sourced Humira®; SB5
Biological: EU sourced Humira®
  Arms: SB5; US sourced Humira®
Biological: US sourced Humira®
  Arms: EU sourced Humira®; US sourced Humira®

SUMMARY:
The purpose of this study is to compare the pharmacokinetics, safety, tolerability, and immunogenicity of SB5 and Humira (EU sourced Humira® and US sourced Humira®) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Have a body mass index between 20.0 and 29.9 kg/m², inclusive.

Exclusion Criteria:

* History and/or current presence of clinical significant atopic allergy, hypersensitivity or allergic reactions, also including known or suspected clinically relevant drug hypersensitivity to any components of the test and reference investigational product formulation or comparable drugs
* Active or latent Tuberculosis or who have a history of Tuberculosis
* History of invasive systemic fungal infections or other opportunistic infections
* Systemic or local infection, a known risk for developing sepsis and/or known active inflammatory process
* Serious infection associated with hospitalisation and/or which required intravenous antibiotics
* History of and/or current cardiac disease
* Have received live vaccine(s) within 4 weeks prior to Screening or who will require live vaccine(s) between Screening and the final study visit
* Intake medication with a half-life > 24 h within 4 weeks or 10 half-lives of the medication prior to investigational product administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Investigational Site, Berlin, Germany

REFERENCES:
- [Derived] Huizinga TWJ, Torii Y, Muniz R. Adalimumab Biosimilars in the Treatment of Rheumatoid Arthritis: A Systematic Review of the Evidence for Biosimilarity. Rheumatol Ther. 2021 Mar;8(1):41-61. doi: 10.1007/s40744-020-00259-8. Epub 2020 Dec 1. PMID 33263165

RESULTS

PARTICIPANT FLOW:
Groups:
- SB5 (Proposed Adalimumab Biosimilar): SB5, single dose of 40 mg via subcutaneous injection (study drug)
  SB5
  EU sourced Humira®
- EU Sourced Humira®: EU sourced Humira®, single dose of 40 mg via subcutaneous injection (reference drug)
  SB5
  US sourced Humira®
- US Sourced Humira®: US sourced Humira®, single dose of 40 mg via subcutaneous injection (reference drug)
  EU sourced Humira®
  US sourced Humira®
Period: Overall Study
Arm/Group | SB5 (Proposed Adalimumab Biosimilar) | EU Sourced Humira® | US Sourced Humira®
Started | 63 | 63 | 63
Completed | 63 | 63 | 63
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB5 (Proposed Adalimumab Biosimilar) | EU Sourced Humira® | US Sourced Humira® | Total
Number analyzed (Participants) | 63 | 63 | 63 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (9.55) | 40.2 (11.06) | 40.0 (10.94) | 39.5 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 6 | 15
  Male | 59 | 58 | 57 | 174
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 61 | 60 | 62 | 183
  Race: Asian | 0 | 2 | 0 | 2
  Race: Black or African American | 2 | 0 | 1 | 3
  Race: Mixed | 0 | 1 | 0 | 1
Height (cm) [Mean (Standard Deviation); unit: cm] | 177.8 (6.72) | 177.5 (6.34) | 177.0 (6.68) | 177.4 (6.56)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 78.83 (7.163) | 78.19 (6.388) | 78.12 (6.458) | 78.38 (6.651)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 24.98 (2.301) | 24.82 (1.823) | 24.97 (1.959) | 24.93 (2.028)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: pre-dose (0 h) and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 336, 504, 672, 1008, 1344, and 1680 h post-dose
Time Frame: 0 to 1680 hours post-dose
Population: Overall number of participans Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Mean (Standard Deviation); unit: μg·h/mL
Arm/Group | SB5 (Proposed Adalimumab Biosimilar) | EU Sourced Humira® | US Sourced Humira®
Number analyzed (Participants) | 53 | 61 | 57
μg·h/mL | 2405.6 (825.93) | 2435.5 (915.66) | 2422.6 (957.00)

2. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: pre-dose (0 h) and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 336, 504, 672, 1008, 1344, and 1680 h post-dose
Time Frame: pre-dose (0 h) and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 336, 504, 672, 1008, 1344, and 1680 h post-dose
Population: Overall number of participans Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | SB5 (Proposed Adalimumab Biosimilar) | EU Sourced Humira® | US Sourced Humira®
Number analyzed (Participants) | 53 | 61 | 57
μg/mL | 3.365 (0.9796) | 3.548 (1.1811) | 3.488 (1.0779)

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Description: pre-dose (0 h) and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 336, 504, 672, 1008, 1344, and 1680 h post-dose
Time Frame: 0 to 1680 hours post-dose
Population: Overall number of participans Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Mean (Standard Deviation); unit: μg·h/mL
Arm/Group | SB5 (Proposed Adalimumab Biosimilar) | EU Sourced Humira® | US Sourced Humira®
Number analyzed (Participants) | 53 | 61 | 57
μg·h/mL | 2125.7 (689.92) | 2096.0 (791.28) | 2101.9 (795.56)

4. Secondary Outcome: Time to Cmax (Tmax)
Description: pre-dose (0 h) and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 336, 504, 672, 1008, 1344, and 1680 h post-dose
Time Frame: pre-dose (0 h) and at 6, 12, 24, 48, 72, 96, 108, 120, 132, 144, 168, 336, 504, 672, 1008, 1344, and 1680 h post-dose
Population: Overall number of participans Analyzed equals to number of subjects who contributed to summary statistics.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SB5 (Proposed Adalimumab Biosimilar) | EU Sourced Humira® | US Sourced Humira®
Number analyzed (Participants) | 53 | 61 | 57
h | 165.962 (89.2503) | 149.715 (76.6421) | 166.456 (79.9227)

ADVERSE EVENTS:
Time Frame: The PK, safety, tolerability, and immunogenicity assessments were performed for maximum 10 weeks after single-dose administration of SB5, EU sourced Humira®, or US sourced Humira®.
Arm/Group | SB5 (Proposed Adalimumab Biosimilar) | EU Sourced Humira® | US Sourced Humira®
Serious Adverse Events (participants affected / at risk) | 1/63 | 0/63 | 1/63
Other Adverse Events (participants affected / at risk) | 29/63 | 17/63 | 25/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB5 (Proposed Adalimumab Biosimilar) (N=63) | EU Sourced Humira® (N=63) | US Sourced Humira® (N=63)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB5 (Proposed Adalimumab Biosimilar) (N=63) | EU Sourced Humira® (N=63) | US Sourced Humira® (N=63)
Nasopharyngitis (Infections and infestations) | 12 (12) | 8 (8) | 11 (11)
Oral herpes (Infections and infestations) | 4 (4) | 1 (1) | 4 (4)
Rhinitis (Infections and infestations) | 2 (2) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 11 (15) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes